CLINICAL TRIAL: NCT06197035
Title: Coping and Caring for Families With Babies With Down Syndrome. A Family-centered Intervention
Brief Title: The Coping With and Caring for Infants With Special Needs Intervention in Down Syndrome Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USeville-EPINTO
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Down Syndrome; Family; Physical Disability
MeSH Terms: conditions — Down Syndrome | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Two intervention groups, a group with COPCA intervention and a group with standard physiotherapy
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPCA (Coping With and Caring for Infants With Special Needs) Intervention (Experimental): The intervention will be delivered by COPCA coaches who follow the programme's theoretical and practical principles. Caregivers learnt how to stimulate their infant's development by challenging their motor behaviour with trial and error experiences.
  This aim to empower the caregivers' competencies to stimulate the infant's daily development, by increasing their motor repertoire.
  and enhancing their capacity to adapt movements to situations.
  Interventions: Procedure: Coping With and Caring for Infants With Special Needs
- Standard physiotherapy (Active Comparator): Standard care will be based on what paediatric physiotherapists generally assume to be useful to promote the development of infants with special needs. Standard care is heterogeneous and eclectic, uses parent training and often includes components of neurodevelopmental treatment with hands-on techniques.
  Interventions: Procedure: Standard Physiotherapy

INTERVENTIONS:
Procedure: Coping With and Caring for Infants With Special Needs — The early intervention programme for infants and young children focuses on the active inclusion of the whole family. The coaching of parents is a central component. Parents learn how they can independently and optimally support their child's development as part of the child's everyday life. The programme was developed at the beginning of the 2000s in the Netherlands by child physiotherapist Tineke Dirks and professor of developmental neurology Mijna Hadders-Algra.
  Arms: COPCA (Coping With and Caring for Infants With Special Needs) Intervention
Procedure: Standard Physiotherapy — Pediatric physiotherapy techniques aimed at improving the development of the baby and young child from manual therapy tools, or baby management.
  Arms: Standard physiotherapy

SUMMARY:
The objective is to compare the impact of standard infant physical therapy and the family-centered program, Coping with and Caring for Infants with Special Needs (COPCA), on infants born with Down syndrome. This is a randomized controlled trial that will be carried out in the patients' homes and outpatient settings in Spain between January 2024 and March 2024. An evaluation battery will be used that includes child and family outcomes and video analysis of therapy sessions.

The Infant Motor profile will be the primary outcome instrument.

ELIGIBILITY:
Inclusion Criteria:

* Babies with Down syndrome
* Families involved in Pediatric Physical Therapy

Exclusion Criteria:

* Other associated developmental disorders
* To not speak Spanish
* Do not sign informed consent

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Motor Development | 3-6-18 months.
  INFANT MOTOR PROFILE Results achieved between the 10% and 90% percentiles indicate adequate motor development. Results between the 5% and 10% percentiles indicate a risk for delays or problems in gross motor development.

SECONDARY OUTCOMES:
Family empowerment | 3-6-18 months
  Family Empowerment Scale
  There are 28 items to be answered by the family with these options:
  1= Strongly Agree' 2= Agree' 3= Disagree' 4= Strongly Disagree. The higher the score, the greater the empowerment.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pinero-Pinto, PhD, Study Director — University of Seville
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
The publication of the results of this research is planned.
Supporting Information: Study Protocol
Time Frame: In 6 months
Access Criteria: Asking t the investigator